CLINICAL TRIAL: NCT05899816
Title: A Phase 3, 24-week, Randomized, Placebo-controlled, Double-blind Study to Assess the Effect of Rocatinlimab on Vaccine Antibody Response in Adult Subjects With Moderate-to-severe Atopic Dermatitis (AD) (ROCKET - VOYAGER)
Brief Title: A Study Assessing Rocatinlimab on Vaccine Antibody Response in Moderate-to-severe Atopic Dermatitis (AD) (ROCKET - VOYAGER)
Acronym: ROCKET-VOYAGER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20210158
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis; Moderate-to-severe Atopic Dermatitis
Keywords: Moderate-to-severe Atopic Dermatitis; AD; Rocatinlimab
MeSH Terms: conditions — Dermatitis, Atopic | interventions — KHK4083

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rocatinlimab (Experimental): Rocatinlimab every 4 weeks (Q4W) for 24 weeks with a loading dose at Week 2.
  Interventions: Drug: Rocatinlimab
- Placebo (Placebo Comparator): Placebo every 4 weeks (Q4W) for 24 weeks with a loading dose at Week 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rocatinlimab — Subcutaneous (SC) injection
  Other Names: AMG 451; KHK4083
  Arms: Rocatinlimab
Drug: Placebo — SC injection
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to:

* estimate vaccine response in rocatinlimab group vs placebo group, assessed using antibody anti-tetanus response at Week 24
* estimate vaccine response in rocatinlimab group vs placebo group, assessed using antibody anti-meningococcal response at Week 24

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years to 54 years with a diagnosis of AD according to the American Academy of Dermatology (AAD) Consensus Criteria (2014) present for at least 12 months
* History of inadequate response to topical corticosteroids (TCS) of medium, high, or higher potency (with or without topical calcineurin inhibitors)
* Subjects with previous systemic treatment for AD are also considered as inadequate responders to topical treatments and are potentially eligible to be included in the study after appropriate washout.
* Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD) score ≥ 3

Exclusion Criteria:

* Treatment with a biologic product within 12 weeks or 5 half-lives, whichever is longer, prior to Day 1
* Treatment with any of the following medications or therapies within 4 weeks or 5 half-lives, whichever is longer, prior to Day 1:

  * Systemic corticosteroids
  * Systemic immunosuppressants
  * Phototherapy
  * Janus kinase inhibitors
* Treatment with any of the following medications or therapies within 1 week, prior to Day 1:

  * TCS of any potency
  * Topical calcineurin inhibitors (TCI)
  * Topical Phosphodiesterase-4 inhibitors (PDE4)
  * Other topical immunosuppressive agents
  * Combination topical agents containing a corticosteroid or calcineurin inhibiting component, PDE4 inhibitors, or other topical immunosuppressive agents
* Treatment with live virus including live attenuated vaccination 12 weeks prior to day 1 pre-randomization.
* Treatment with any meningococcal vaccine within 1 year prior to screening, or treatment with any tetanus-, diphtheria-, or pertussis containing vaccine within 5 years prior to screening

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a Positive Anti-tetanus Response | Week 20 to week 24
Number of Participants with a Positive Anti-meningococcal Response | Week 20 to week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (85):
- United States (72):
  - Affiliated Dermatology, Scottsdale, Arizona
  - Center for Dermatology and Plastic Surgery, Scottsdale, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Medical Advancement Centers of Arizona, Tempe, Arizona
  - Little Rock Allergy and Asthma Clinical Research Center, Little Rock, Arkansas
  - Kern Research Inc, Bakersfield, California
  - Hope Clinical Research LLC, Canoga Park, California
  - Doc1 Healthcare Systems, Chino, California
  - 310 Clinical Research, Inglewood, California
  - Chemidox Clinical Trials Incorporated, Lancaster, California
  - Long Beach Research Institute, Long Beach, California
  - University of California Los Angeles, Los Angeles, California
  - Wallace Medical Group Inc, Los Angeles, California
  - West Los Angeles Clinical Trials, Los Angeles, California
  - Northridge Clinical Trials, Northridge, California
  - Havana Research Institute Inc, Pasadena, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Integrative Skin Science and Research, Sacramento, California
  - Wake Research Medical Center for Clinical Research, San Diego, California
  - Cura Clinical Research, Sherman Oaks, California
  - Wolverine Clinical Trials, Tustin, California
  - Alliance for Multispecialty Research, Coral Gables, Florida
  - Life Clinical Trials, Coral Springs, Florida
  - AllerVie Clinical Research- Destin, Destin, Florida
  - D and H Doral Research Centers, Doral, Florida
  - Saint Jude Clinical Research, Doral, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Nexus Clinical Research, Homestead, Florida
  - D and H National Research Centers, Miami, Florida
  - Gold Coast Health Research Center, Miami, Florida
  - Anchor Medical Research, Miami, Florida
  - Meridian International Research, Miami Gardens, Florida
  - AllerVie Clinical Research- Ocala, Ocala, Florida
  - D and H Tamarac Research Centers, Tamarac, Florida
  - Hamilton Research, LLC, Alpharetta, Georgia
  - Divine Dermatology and Aesthetics, Atlanta, Georgia
  - MetroDerm / Atlanta Center for Clinical Research, LLC, Atlanta, Georgia
  - First Georgia Physicians Group, Fayetteville, Georgia
  - Dermatologic Surgery Specialists, Macon, Georgia
  - McIntosh Clinic PC, Thomasville, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - Dermatology and Skin Cancer Center Leawood, Leawood, Kansas
  - Visage Dermatology and Aesthetic Center, Largo, Maryland
  - ActivMed Practices and Research, LLC, Methuen, Massachusetts
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - The Derm Institute of West Michigan, Caledonia, Michigan
  - Excel Clinical Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Pioneer Clinical Research New York, New York, New York
  - Rochester Clinical Research Inc, Rochester, New York
  - Hickory Dermatology Research Center, Hickory, North Carolina
  - Tryon Medical Partners, Matthews, North Carolina
  - The Skin Surgery Center, Winston-Salem, North Carolina
  - Apex Clinical Research Center LLC, Mayfield Heights, Ohio
  - Dermatologist of Central States Clinical Research - Springfield, Springfield, Ohio
  - Epic Medical Research - Oklahoma, Chickasha, Oklahoma
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Dermatology Research Center of Oklahoma, PLLC, Tulsa, Oklahoma
  - Velocity Clinical Research Inc, Medford, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Cumberland Skin Center, Hermitage, Tennessee
  - MedCare Pharma - Houston, Houston, Texas
  - sms Clinical Research Limited Liability Company, Mesquite, Texas
  - Stryde Research - Epiphany Dermatology, Southlake, Texas
  - Tranquil Clinical Research, Webster, Texas
  - Cope Family Medicine, Bountiful, Utah
  - Tanner Clinic, Murray, Utah
- Canada (13):
  - Skin Physicians Dermatology, Edmonton, Alberta
  - Interior Dermatology Centre, Kelowna, British Columbia
  - Karma Clinical Trials, St. John's, Newfoundland and Labrador
  - Skincare Studio, St. John's, Newfoundland and Labrador
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - York Dermatology Centre, Richmond Hill, Ontario
  - FACET Dermatology, Toronto, Ontario
  - Evidence Based Medical Educator Inc, Toronto, Ontario
  - DermAtelier Clinical Research Incorporated, Toronto, Ontario
  - Clinique de Dermatologie Rosemont, Montreal, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Sima recherche, Verdun, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Guttman-Yassky E, Simpson E, Bissonnette R, Eichenfield LF, Kabashima K, Luna PC, Hercogova JT, Spelman L, Worm M, Esfandiari E, Arai T, Mano H, Charuworn P, Wang A, Kricorian G. ROCKET: a phase 3 program evaluating the efficacy and safety of rocatinlimab in moderate-to-severe atopic dermatitis. Immunotherapy. 2025 Feb;17(2):83-94. doi: 10.1080/1750743X.2025.2464528. Epub 2025 Feb 26. PMID 40012373
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com